CLINICAL TRIAL: NCT02337413
Title: A Controlled Randomized, Physician Blinded Study to Assess Isolated Uro-therapy vs. Urotherapy With Constipation Treatment for Patients With Moderate-severe Monosymptomatic Nocturnal Enuresis (MNE) Not Meeting ROME-III Constipation Criteria
Brief Title: Urotherapy vs. Urotherapy With Constipation Treatment for Nocturnal Enuresis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Changes in departmental staff have led to a cut in research alotments.
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Noam Zevit, Pediatric Gastroenterologist, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: rmc130342ctil
Record Dates: First submitted 2015-01-01; First posted 2015-01-13 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Nocturnal Enuresis
Keywords: Constipation
MeSH Terms: conditions — Nocturnal Enuresis; Constipation | interventions — polyethylene glycol 3350

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urotherapy + Constipation Treatment (Active Comparator): This group will be treated with standard behavioral urotherapy in addition to receiving active stool softening with PEG3350 and standard constipation instruction.
  Interventions: Drug: Polyethylene glycol 3350; Behavioral: Constipation behavioral therapy; Behavioral: Urotherapy
- Urothearpy alone (Other): This group will receive standard behavioral urotherapy alone
  Interventions: Behavioral: Urotherapy

INTERVENTIONS:
Drug: Polyethylene glycol 3350 — Patients will initially receive three days of high dose PEG3350 treatment (1.5gr/kg up to 100gr maximum) and then will be stepped down to 0.8gr/kg subsequently and tapered accoriding to stool consistency and frequency.
  Other Names: Normalax
  Arms: Urotherapy + Constipation Treatment
Behavioral: Constipation behavioral therapy — Patients in the active group will receive dietary instruction as to fiber content, as well as behavioral therapy including active sitting on the toilet to attempt defaction following meals.
  Arms: Urotherapy + Constipation Treatment
Behavioral: Urotherapy — Patients will be guided for appropriate drinking and toilet habits, and will start with timed voiding.

SUMMARY:
Constipation treatment has been found to ameliorate symptoms in some patients with nocturnal enuresis (bed wetting at night). This study aims to explore if treatment of patients without overt constipation (As defined by the ROME III criteria) will also respond to stool softening and GI behavioral therapy with reduction of their urinary tract symptoms when added to standard urotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 5-17 years at time of signing of informed consent.
2. MNE as defined by ≥3 wet nights/week without daytime incontinence
3. Do not meet Rome III criteria for functional constipation

Exclusion Criteria:

1. Inability to provide signed informed consent.
2. Inability to comply with the study protocol.
3. Neurogenic bladder
4. Attention Deficit Disorder (ADD or ADHD) on medical treatment.
5. Known significant sacral, perineal, or other congenital or surgical defect.
6. Known orthopedic/neurological disease which may affect urinary continence, cause constipation, or affect reading of abdominal x-rays. (e.g. spastic cerebral palsy, severe scoliosis)
7. Patient taking medicinal drugs which can cause urinary incontinence or constipation.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with complete (no nocturnal enuresis) or partial (A decease in nocturnal enuresis episodes of 50% or more) response at week 14 | 14 weeks
  Proportion of patients with uro-therapy + constipation treatment with complete (No nocturnal enuresis) or partial (A decease in nocturnal enuresis episodes of 50% or more) response in comparison to the isolated urotherapy group.

SECONDARY OUTCOMES:
Number of participants with complete (no nocturnal enuresis) or Partial (A decease in nocturnal enuresis episodes of 50% or more) response of enuresis to treatment in patient subgroups with fecal loading compared to those without fecal loading. | 14 weeks
  Complete (no nocturnal enuresis) or Partial (A decease in nocturnal enuresis episodes of 50% or more) response to therapy in those with radiological evidence of fecal loading on enrollment abdominal x-ray (as defined by rectal/pelvic outlet ratio, Leech score, and Barr score) compared to those who did not in the intervention group and the urotherapy group.
Number of participants with sustained complete (no nocturnal enuresis) or partial (A decease in nocturnal enuresis episodes of 50% or more) response 12 weeks after the end of the intervention. | 26 weeks
  Sustained complete (no nocturnal enuresis) or Partial (A decease in nocturnal enuresis episodes of 50% or more) response at 26 weeks.
Number of participants with adverse effects | 14 weeks
  Adverse effects of interventions as reported by patients/care givers during visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Gastroenterology, Nutrition and Liver Diseases; Schneider Children's Medical Center of Israel, Petah Tikva, Israel

REFERENCES:
- [Background] Hodges SJ, Anthony EY. Occult megarectum--a commonly unrecognized cause of enuresis. Urology. 2012 Feb;79(2):421-4. doi: 10.1016/j.urology.2011.10.015. Epub 2011 Dec 14. PMID 22173180